CLINICAL TRIAL: NCT03273608
Title: Superselective Drug-Eluting Chemoembolization in Unresectable Intermediate and Advanced HCC Patients: Safety & Efficacy Registry in Taiwan (SUPER- Taiwan)
Brief Title: Observation Study: Superselective Drug-Eluting Chemoembolization in Unresectable Intermediate and Advanced HCC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Taiwan University Hospital (Other); Tri-Service General Hospital (Other); China Medical University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, vghtpe user, Professor Yi-Hsiang Huang, Taipei Veterans General Hospital, Taiwan
Other Study IDs: HEPA-Taiwan-001
Record Dates: First submitted 2017-08-04; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Advanced HCC; Unresectable; deTACE; HepaSphere
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this multicenter registry is to gather the safety, efficacy and survival data in intermediate and advanced HCC patients treated drug-eluting microsphere in Taiwan in order to provide clinical evidence in HCC management to physicians in the region, and to support the application of deTACE in treating advanced HCC patients.

DETAILED DESCRIPTION:
The purpose of this multicenter registry is to gather the safety, efficacy and survival data in intermediate and advanced HCC patients treated drug-eluting microsphere in Taiwan in order to provide clinical evidence on deTACE in HCC management to physicians in the region, and to support the application of in treating advanced HCC patients.

1. Primary Objective:

   To collect 1-year overall survival of chemoembolization with drug-eluting microsphere in intermediate and advanced HCC patients in Taiwan.
2. Secondary Objectives:

   1. To evaluate the overall tumor response of chemoembolization with drug-eluting microsphere in intermediate and advanced HCC patients. The tumor response is according to Modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.
   2. To evaluate the local tumor response (in the tumor(s) treated with drug-eluting microsphere) by chemoembolization with drug-eluting microsphere in intermediate and advanced HCC patients.
   3. To evaluate the safety profile of chemoembolization with drug-eluting microsphere in intermediate and advanced HCC patients.
3. Exploratory Objectives:

   1. To evaluate the downstaging and downsizing potential of chemoembolization with drug-eluting microsphere in intermediate and advanced HCC patients to within Milan Criteria and to within Resection margin.
   2. To collect time-to-progression (TTP) and progress-free-survival (PFS) data of chemoembolization with drug-eluting microsphere in intermediate and advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:Patients must meet all of the following inclusion criteria in order to be entered into the study:

* Age 20 or older.
* Patient has signed informed consent.
* Patient must have a diagnosis of hepatocellular cancer confirmed by AASLD and at least one of the following method:

  * Magnetic resonance imaging (MRI) with early enhancement and delayed enhancement washout of at least one solid liver lesion > 1 cm.
  * Contrast enhanced computed tomography (CT) with early enhancement and delayed enhancement washout of at least one solid liver lesion > 1 cm.
  * Histological confirmation is required for lesions with inconclusive features.
* Patient must not be suitable for treatment by resection or percutaneous ablation at time of study entry.

  * Patients not suitable for ablation due to lesion location may be enrolled.
  * Patients with HCC recurrence but not suitable for resection or ablation maybe enrolled.
* Patient MUST be with either BCLC stage B OR C, and meet the following criteria:

  * Stage Child-Pugh A or B AND
  * Performance status ECOG ≤ 1 WITH Vascular Invasion or WITHOUT Vascular invasion.
* Patient has a life expectancy of at least 6 months.

Exclusion Criteria:If patients meet any of the following criteria they may not be entered into the study:

* Current or previous treatment with chemo- or radiation therapy or sorafenib or drug-eluting chemoembolization (deTACE).
* Patients with concurrent cancer except non-melanomatous skin cancer.
* Female patients who are pregnant, breastfeeding, or premenopausal and not using an effective method of contraceptive.
* Performance status ECOG > 1.
* Child-Pugh Class C.
* Occlusive tumor thrombus to the main portal trunk.
* Active gastrointestinal bleeding.
* Evidence of uncorrectable bleeding diathesis.
* Extra-Hepatic spread of the HCC.
* Encephalopathy not adequately controlled medically.
* Presence of ascites not controlled medically.
* Any contraindication for MRI/ CT (eg. metallic implants).
* Allergy to contrast media that cannot be managed with prophylaxis.
* Any contraindication to arteriography.
* Any contraindication for doxorubicin administration.
* Any contraindication for hepatic embolization. Porto-systemic shunt, or an arteriovenous shunt that cannot be adequately closed prior to chemoembolization. Hepatofugal blood flow. Serum creatinine > 2mg/dL. Other condition deemed exclusionary by physician. Uncorrectable impaired clotting.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Superselective Drug-Eluting Chemoembolization in Unresectable Intermediate and Advanced HCC Patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-09-14 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  To define all participants from the day of the first HepaSphere Treatment until end of study or death is reported, whichever comes first.

SECONDARY OUTCOMES:
Tumor Response | 1 year
  Tumor response will be assessed using modified Response Evaluation Criteria In Solid Tumors (mRECIST) criteria to evaluate tumor necrosis under CT/ MRI and will be presented as %.
Adverse Event (AE) | 1 year
  Adverse event will be accessed according to CTCAE 4.0 after treatments until end of study or death.

OTHER OUTCOMES:
Exploratory Objectives, Time-To-Progression (TTP) | 1 year
  To define all participants from the day of the first HepaSphere Treatment until tumor progression or death is first reported, whichever comes first.
Exploratory Objectives, Downstaging | 1 year
  Tumor staging will be accessed according to BCLC staging system and Milan criteria, and will be reviewed at follow-up until end of study or death.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsiang Huang, M.D. Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan